CLINICAL TRIAL: NCT06536465
Title: A Phase 2 Clinical Study of REC-3964 in Adults for the Reduction of Recurrent Clostridioides Difficile Infection (CDI)
Brief Title: The Clostridioides Difficile Trial of REC-3964
Acronym: ALDER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to sponsor decision. This decision was not related to safety concerns.
Sponsor: Recursion Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-3964-201
Record Dates: First submitted 2024-07-15; First posted 2024-08-05 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Clostridioides Difficile Infection
Keywords: Cdiff Infection; Clostridiodes difficile infection; Cdiff
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- REC-3964 High-dose (Experimental): Participants will receive 500 mg REC-3964 q12h REC-3964 250 mg capsules
  Interventions: Drug: REC-3964
- REC-3964 Low-dose (Experimental): Participants will receive 250 mg REC-3964 q12h REC-3964 250 mg capsules
  Interventions: Drug: REC-3964
- Observation (No Intervention): Participants will undergo watchful waiting

INTERVENTIONS:
Drug: REC-3964 — REC-3964 given at a dose of either 500 mg q12h or 250 mg q12h
  Arms: REC-3964 High-dose; REC-3964 Low-dose

SUMMARY:
This is a multi-center, open-label study to investigate the safety, tolerability, pharmacokinetics (PK) and efficacy of REC-3964 (doses of either 250 mg or 500 mg PO every 12 hours) for the reduction of Clostridioides difficile infection (CDI).

DETAILED DESCRIPTION:
Study was terminated due to sponsor decision. This decision was not related to safety concerns.

ELIGIBILITY:
Key Inclusion Criteria:

* Be 18 years of age or older with Clostridioides difficile infection (CDI) diarrhea associated with a positive stool test for C. difficile toxin[s] prior to the preceding curative treatment.
* The CDI episode, severe or otherwise, must have resolved after receiving vancomycin with a standard duration of treatment. The participant must be randomized within 2 days of completing the preceding curative treatment.
* Have high risk for rCDI (a recurrent CDI episode within the last 6 months, age ≥65 years, immunocompromised state, or severe CDI with resolution prior to enrollment into the study).

Key Exclusion Criteria:

* Have an active, symptomatic, chronic diarrheal illness from other causes, such as ulcerative colitis or Crohn's disease.
* Diarrhea that requires on-study treatment with agents that would confound the interpretation of the study results.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GANJ - Toms River - Ocean Family Gastroenterology, Toms River, New Jersey
  - Southern Star Research Institute, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to early study termination, only 3 participants were enrolled.
Groups:
- REC-3964 250 mg: Participants received REC-3964 given at a dose 250 milligrams (mg) every 12 hours (q12h).
- REC-3964 500 mg: Participants received REC-3964 given at a dose of 500 mg q12h.
- Observation: Participants underwent watchful waiting. No treatment was administered.
Period: Overall Study
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
Started | 1 | 1 | 1
Completed | 1 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants. Due to the small sample size, data were not reported for participant confidentiality reasons.
Groups:
- REC-3964 250 mg: Participants received REC-3964 given at a dose 250 mg q12h.
- Total: Total of all reporting groups
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Due to the small sample size, data was not reported for participant confidentiality reasons.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to the small sample size, data was not reported for participant confidentiality reasons.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the small sample size, data was not reported for participant confidentiality reasons.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to the small sample size, data was not reported for participant confidentiality reasons.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Survival Without Recurrence or Requirement for Additional Clostridioides Difficile Infection (CDI) Treatment
Description: Recurrent CDI was defined as a new episode of CDI associated with a new positive Clostridioides difficile stool toxin or requirement for additional CDI treatment during the 8-week Follow-up Period after cure of preceding CDI with initial curative treatment.
Time Frame: 8 weeks
Population: All randomized participants who received at least 1 dose of REC-3964 intervention or who were followed-up on in the Observational arm.
Measure: Count of Participants; unit: Participants
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
Number analyzed (Participants) | 1 | 1 | 1
Participants | 1 | 1 | 1

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product.
Time Frame: Up to 8 weeks
Population: All randomized participants who received at least 1 dose of REC-3964 intervention or who were followed-up on in the Observation arm.
Measure: Count of Participants; unit: Participants
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
Number analyzed (Participants) | 1 | 1 | 1
Participants | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Related TEAEs
Description: A TEAE was the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An Investigator who was qualified in medicine determined relationship to the study drug for each AE (unrelated or related). The Investigator decided whether, in his or her medical judgment, if there was a reasonable biological possibility that the event may have been caused by the study drug.
Time Frame: Up to 8 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
Number analyzed (Participants) | 1 | 1 | 1
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Serious TEAEs
Description: A TEAE was the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. A Serious TEAE was defined as results in death, immediately life-threatening, requires in-participant hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity in conducting activities of daily living for at least 28 days, results in a congenital abnormality or birth defect, or an important medical event that may jeopardize the participant or may require medical intervention.
Time Frame: Up to 8 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
Number analyzed (Participants) | 1 | 1 | 1
Participants | 0 | 0 | 0

5. Primary Outcome: Number of Participants With TEAEs Leading to Study Drug Discontinuation
Description: as for outcome 2
Time Frame: Up to 8 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
Number analyzed (Participants) | 1 | 1 | 1
Participants | 0 | 0 | 0

6. Secondary Outcome: Rate of Recurrent Clostridioides Difficile Infection (rCDI)
Description: Recurrent CDI was defined as a new episode of CDI associated with a new positive Clostridioides difficile stool toxin within 8 weeks of the cessation of initial curative treatment. The number of unformed [types 5-7 on the Bristol stool scale] bowel movements per day were recorded by the participant in the stool diary in order to identify a new episode of diarrhea. All new episodes of diarrhea were tested for toxigenic Clostridioides difficile to confirm CDI recurrence.
  The rate of rCDI was defined as the proportion of participants who had the Clostridioides difficile recurrence among randomized participants.
Time Frame: 8 weeks
Population: Data for this outcome measure was not summarized since there was only 1 participant in each treatment arm.
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Time to Recurrence of rCDI
Description: Recurrent CDI was defined as a new episode of CDI associated with a new positive Clostridioides difficile stool toxin within 8 weeks of the cessation of initial curative treatment. The number of unformed [types 5-7 on the Bristol stool scale] bowel movements per day were recorded by the participant in the stool diary in order to identify a new episode of diarrhea. All new episodes of diarrhea were tested for toxigenic Clostridioides difficile to confirm CDI recurrence. Time to recurrence of rCDI was to be assessed using Kaplan-Meier estimation.
Time Frame: Up to 8 weeks
Population: Data for this outcome measure could not be estimated since no recurrence events occurred during this study.
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Severe rCDI
Description: Recurrent CDI was defined as a new episode of CDI associated with a new positive Clostridioides difficile stool toxin within 8 weeks of the cessation of initial curative treatment. The number of unformed [types 5-7 on the Bristol stool scale] bowel movements per day were recorded by the participant in the stool diary in order to identify a new episode of diarrhea. All new episodes of diarrhea were tested for toxigenic Clostridioides difficile to confirm CDI recurrence. Severe CDI was defined as CDI with white blood cell count >15,000 cells/milliliter and/or serum creatinine ≥1.5 milligram/deciliter.
Time Frame: Up to 8 weeks
Population: Data for this outcome measure was not assessed since no recurrence events occurred.
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With rCDI Who Had Associated Hospital Admissions
Description: Recurrent CDI was defined as a new episode of CDI associated with a new positive Clostridioides difficile stool toxin within 8 weeks of the cessation of initial curative treatment. The number of unformed [types 5-7 on the Bristol stool scale] bowel movements per day were recorded by the participant in the stool diary in order to identify a new episode of diarrhea. All new episodes of diarrhea were tested for toxigenic Clostridioides difficile to confirm CDI recurrence.
Time Frame: Up to 8 weeks
Population: Data for this outcome measure was not assessed since no recurrence events occurred.
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of REC-3964
Time Frame: Pre-dose, 1 hour, 3 hours, and 6 hours post morning dose on Day 1 and Day 15
Population: Data for this outcome measure was not summarized since there was only 1 participant in each treatment arm.
Arm/Group | REC-3964 250 mg | REC-3964 500 mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of REC-3964
Time Frame: Pre-dose, 1 hour, 3 hours, and 6 hours post morning dose on the Day 1 and Day 15
Population: Data for this outcome measure was not summarized since there was only 1 participant in each treatment arm.
Arm/Group | REC-3964 250 mg | REC-3964 500 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Trough Plasma Concentration (Ctrough) of REC-3964
Time Frame: Pre-dose on Day 15
Population: Data for this outcome measure was not summarized since there was only 1 participant in each treatment arm.
Arm/Group | REC-3964 250 mg | REC-3964 500 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: All randomized participants who received at least 1 dose of REC-3964 intervention or who were followed-up on in the Observation arm.
  AEs occurring in participants randomized to observation were recorded up to 28 days after the participant's last day in the Observation arm.
Arm/Group | REC-3964 250 mg | REC-3964 500 mg | Observation
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | REC-3964 250 mg (N=1) | REC-3964 500 mg (N=1) | Observation (N=1)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, only 3 participants were enrolled. Data are limited due to the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT06536465/Prot_SAP_000.pdf